CLINICAL TRIAL: NCT03946670
Title: A Randomized, Double-blind, Placebo-controlled Phase II Multi-center Study of Intravenous MBG453 Added to Hypomethylating Agents in Adult Subjects With Intermediate, High or Very High Risk Myelodysplastic Syndrome (MDS) as Per IPSS-R Criteria
Brief Title: A Study of MBG453 in Combination With Hypomethylating Agents in Subjects With IPSS-R Intermediate, High or Very High Risk Myelodysplastic Syndrome (MDS).
Acronym: STIMULUS-MDS1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In December 2023, Novartis decided to terminate the sabatolimab clinical development program early after Phase II (MDS1) and Phase III (MDS2) studies failed to meet their primary objectives. The termination was not due to safety concerns.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMBG453B12201; 2018-004479-11 (EudraCT Number)
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Myelodysplastic Syndromes
Keywords: Sabatolimab; Placebo; Phase II; MBG453; TIM-3; decitabine; azacitidine; myelodysplastic syndrome (MDS)
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — sabatolimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MBG453 + hypomethylating agents (Experimental): Patients are taking MBG453 plus hypomethylating agents
  Interventions: Drug: MBG453; Drug: Hypomethylating agents
- Placebo + hypomethylating agents (Placebo Comparator): Patients are taking placebo plus hypomethylating agents
  Interventions: Drug: Placebo; Drug: Hypomethylating agents

INTERVENTIONS:
Drug: MBG453 — MBG453 is being administered i.v.
  Other Names: Sabatolimab
  Arms: MBG453 + hypomethylating agents
Drug: Placebo — Placebo is being administered i.v.
  Arms: Placebo + hypomethylating agents
Drug: Hypomethylating agents — Decitabine is being administered i.v. Azacitidine is being administered i.v or s.c.

SUMMARY:
This Phase II was a multicenter, randomized, two-arm parallel-group, double-blind, placebo-controlled study of MBG453 or placebo added to hypomethylating agents (azacitidine or decitabine) in adult subjects with IPSS-R intermediate, high or very high risk myelodysplastic syndrome (MDS) not eligible for Hematopoietic Stem Cell Transplant (HSCT) or intensive chemotherapy.

DETAILED DESCRIPTION:
The 2 primary objectives were as follows:

To determine if MBG453 combined with standard HMA therapy improved complete remission in subjects with intermediate, high, or very high risk MDS.

To determine if MBG453 combined with standard HMA therapy improved progression free survival (PFS) in subjects with intermediate, high or very high risk MDS.

This Phase II study was a multicenter, randomized, two-arm parallel-group, double-blind, placebo-controlled study of MBG453 or placebo added to hypomethylating agents (azacitidine or decitabine, as per investigators' choice based on local standard of care (SOC)) in adult subjects with IPSS-R intermediate, high or very high risk MDS not eligible for HSCT or intensive chemotherapy. A total of 127 subjects were randomized in a 1:1 ratio to treatment arms as follows:

* MBG453 400 mg IV Q2W and decitabine or azacitidine
* Placebo IV Q2W and decitabine or azacitidine

The randomization was stratified by 2 stratification factors: a) HMA (decitabine or azacitidine) selected by the investigator as per the local SOC and b) IPSS-R prognostic risk categories (intermediate, high or very high) at randomization. Crossover between treatment arms was not permitted at any time during the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Age ≥ 18 years at the date of signing the informed consent form (ICF)-. Morphologically confirmed diagnosis of a myelodysplastic syndrome (MDS) based on 2016 WHO classification (Arber et al 2016) by investigator assessment with one of the following Prognostic Risk Categories, based on the International Prognostic Scoring System (IPSS-R):

  * Very high
  * High
  * Intermediate with at least ≥ 5% bone marrow blast
* Not eligible at the time of screening, for intensive chemotherapy according to the investigator, based on local standard medical practice and institutional guidelines for treatment decisions
* Not eligible at the time of screening, for hematopoietic stem-cell transplantation (HSCT) according to the investigator, based on local standard medical practice and institutional guidelines for treatment decisions.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Exclusion Criteria:

* Prior exposure to TIM-3 directed therapy at any time. Prior therapy with immune check point inhibitors (e.g. anti-CTLA4, anti-PD-1, anti-PD-L1, or anti-PD-L2), cancer vaccines are allowed except if the drug was administered within 4 months prior to randomization.
* Previous first-line treatment for higher risk MDS with chemotherapy or any other antineoplastic agents including lenalidomide and hypomethylating agent (HMAs) such as decitabine or azacitidine.
* History of severe hypersensitivity reactions to any ingredient of the study treatment (azacitidine, decitabine or MGB453) or their excipients, or to monoclonal antibodies (mAbs).
* Currently using or used within 14 days prior to randomization of systemic, steroid therapy (> 10 mg/day prednisone or equivalent) or any immunosuppressive therapy. Topical, inhaled, nasal, ophthalmic steroids are allowed. Replacement therapy, steroids given in the context of a transfusion are allowed and not considered a form of systemic treatment.
* Investigational treatment for MDS received within 4 weeks prior to randomization. In case of a checkpoint inhibitor: 4 months minimum prior to randomization interval is necessary to allow enrollment.
* Active autoimmune disease requiring systemic therapy (e.g.corticosteroids).
* Live vaccine administered within 30 Days prior to randomization.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (48):
- United States (7):
  - City Of Hope National Med Center, Duarte, California
  - City of Hope National Medical Center Medical Oncology & Therapeutic, Duarte, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - The Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State Comprehensive Cancer Center James Cancer Hospital, Columbus, Ohio
  - Mary Crowley Cancer Research, Dallas, Texas
- Novartis Investigative Site, Vienna, Austria
- Belgium (2):
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Leuven
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Québec, Quebec
- Czechia (2):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Toulouse, France
- Germany (2):
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Berlin
- Greece (3):
  - Novartis Investigative Site, Alexandroupoli
  - Novartis Investigative Site, Larissa
  - Novartis Investigative Site, Pátrai
- Novartis Investigative Site, Hong Kong, Hong Kong
- Hungary (2):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Nyíregyháza
- Italy (5):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
- Japan (9):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Gifu
  - Novartis Investigative Site, Osaka
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Málaga
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Samsun, Atakum
  - Novartis Investigative Site, Köseköy, Kocaeli
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access Criteria: Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Zeidan AM, Ando K, Rauzy O, Turgut M, Wang MC, Cairoli R, Hou HA, Kwong YL, Arnan M, Meers S, Pullarkat V, Santini V, Malek K, Kiertsman F, Niolat J, Ramos PM, Menssen HD, Fenaux P, Miyazaki Y, Platzbecker U. Sabatolimab plus hypomethylating agents in previously untreated patients with higher-risk myelodysplastic syndromes (STIMULUS-MDS1): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Haematol. 2024 Jan;11(1):e38-e50. doi: 10.1016/S2352-3026(23)00333-2. Epub 2023 Dec 5. PMID 38065203
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 47 centers across 17 countries enrolled subjects in this study.
Groups:
- MBG453 + Hypomethylating Agents (HMA): Participants were taking MBG453 plus hypomethylating agents
- Placebo + Hypomethylating Agents (HMA): Participants were taking placebo plus hypomethylating agents
Period: Overall Study
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Started | 65 | 62
Treated | 64 | 61
Not treated | 1 | 1
Discontinued from treatment | 64 | 61
Completed (Completed = Completed treatment) | 0 | 0
Not Completed | 65 | 62
Not completed — Progressive Disease | 34 | 27
Not completed — Adverse Event | 7 | 10
Not completed — Physician Decision | 6 | 5
Not completed — Death | 5 | 8
Not completed — Hematopoietic stem cell transplantation (HSCT) Planned | 5 | 6
Not completed — Subject Decision | 4 | 5
Not completed — Study Terminated By Sponsor | 2 | 0
Not completed — New Therapy For Study Indication | 1 | 0
Not completed — Not Treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized subjects were included in the FAS (intent-to-treat population) Subject data in the FAS were analyzed according to the treatment and stratum they were assigned to when they were randomized. Efficacy.
Groups:
- Total: Total of all reporting groups
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA) | Total
Number analyzed (Participants) | 65 | 62 | 127
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.9 (6.70) | 71.3 (9.64) | 71.6 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 17 | 41
  Male | 41 | 45 | 86
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 44 | 33 | 77
  Asian | 17 | 25 | 42
  Black or African American | 0 | 1 | 1
  Unknown | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate
Description: CR: where the Bone marrow: ≤ 5% blasts with normal maturation of all cell lineages and Peripheral blood: where Hgb ≥ 10 g/dL AND Platelets ≥ 100*109/L AND Neutrophils ≥ 1.0*109/L AND Peripheral blasts 0%.
  Modified response criteria According to International Working Group (IWG) and as per World Health Organization (WHO) criteria for Myelodysplastic syndromes (MDS) as per investigator assessment.
Time Frame: average of 7 months
Population: Full Analysis Set (FAS): All randomized participants were included in the FAS (intent-to-treat population) Participant data in the FAS were analyzed according to the treatment and stratum they were assigned to when they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
Percentage of participants | 21.5 [12.3 to 33.5] | 17.7 [9.2 to 29.5]
Statistical Analysis 1: Comparison: MBG453 + Hypomethylating Agents (HMA) vs Placebo + Hypomethylating Agents (HMA); Test type: Superiority; p = 0.769, Cochran-Mantel-Haenszel; stratified by the randomization stratification factor IPSS-R category

2. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as time from randomization to disease progression (including transformation to acute leukemia per WHO 2016 classification), relapse from CR according to IWG-MDS or death due to any cause, whichever occurs first, as per investigator assessment.
Time Frame: approx. 32 months
Population: Full Analysis Set (FAS): All randomized participants were included in the FAS (intent-to-treat population). Participant data in the FAS were analyzed according to the treatment and stratum they were assigned to when they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
months | 11.07 [7.62 to 17.61] | 8.48 [6.93 to 11.30]
Statistical Analysis 1: Comparison: MBG453 + Hypomethylating Agents (HMA) vs Placebo + Hypomethylating Agents (HMA); Test type: Superiority; p = 0.1022, Log Rank; stratified by the randomization stratification factor IPSS-R category; Cox Proportional Hazard = 0.749, 95% CI 2-sided [0.479 to 1.173]

3. Secondary Outcome: Progression Free Survival (PFS) - Final PFS
Description: PFS isdefined as time from randomization to disease progression (including transformation to acute leukemia per WHO 2016 classification), relapse from CR according to IWG-MDS or death due to any cause. This is an update of the Primary Outcome Measure PFS with data collected after assessment of the primary results.
Time Frame: approx. 48 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
months | 11.07 [7.62 to 16.59] | 8.48 [6.93 to 11.30]
Statistical Analysis 1: Comparison: MBG453 + Hypomethylating Agents (HMA) vs Placebo + Hypomethylating Agents (HMA); Test type: Superiority; Hazard Ratio (HR) = 0.795, 95% CI 2-sided [0.521 to 1.212] — Cox model stratified by IPSS-R score as per IRT

4. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to death due to any cause
Time Frame: approx. 48 months
Population: Full Analysis Set (FAS): All randomized participants were included in the FAS (intent to treat population). Participant data in the FAS were analyzed according to the treatment and stratum they were assigned to when they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
Months | 19.12 [13.90 to 30.03] | 18.00 [13.11 to 25.43]
Statistical Analysis 1: Comparison: MBG453 + Hypomethylating Agents (HMA) vs Placebo + Hypomethylating Agents (HMA); Test type: Superiority; Hazard Ratio (HR) = 0.808, 95% CI 2-sided [0.542 to 1.205] — Cox model stratified by IPSS-R score as per Interactive Response Technology (IRT)

5. Secondary Outcome: Event-free Survival (EFS)
Description: EFS is defined as the time from randomization to lack of reaching complete response (CR) within the first 6 months, relapse from CR or death due to any cause, whichever occurs first. CR and relapse from CR were defined according to International Working Group (IWG) for Myelodysplastic Syndromes (MDS) as per Investigator assessment. For participants not reaching CR within the first 6 months, an EFS event at day 1 was considered.
Time Frame: approx. 48 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
Months | 0.03 [0.0 to NA] — NA: Because the survival curve crossed below 50% almost immediately, leaving no earlier time point to support calculation and remained below 50% afterward, the lower confidence limit was set to 0 and the upper confidence limits could not be estimable. | 0.03 [0.0 to NA] — NA: Because the survival curve crossed below 50% almost immediately, leaving no earlier time point to support calculation and remained below 50% afterward, the lower confidence limit was set to 0 and the upper confidence limits could not be estimable.
Statistical Analysis 1: Comparison: MBG453 + Hypomethylating Agents (HMA) vs Placebo + Hypomethylating Agents (HMA); Test type: Superiority; Hazard Ratio (HR) = 0.890, 95% CI 2-sided [0.589 to 1.343] — Cox model stratified by IPSS-R score as per IRT

6. Secondary Outcome: Leukemia-free Survival (LFS)
Description: LFS is defined as the time from randomization to ≥ 20% blasts in bone marrow/peripheral blood (per World Health Organization (WHO) 2016 classification) or diagnosis of extramedullary acute leukemia or death due to any cause.
Time Frame: approx. 48 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
Months | 16.82 [8.80 to 28.58] | 13.63 [9.82 to 21.16]
Statistical Analysis 1: Comparison: MBG453 + Hypomethylating Agents (HMA) vs Placebo + Hypomethylating Agents (HMA); Test type: Superiority; Hazard Ratio (HR) = 0.906, 95% CI 2-sided [0.570 to 1.440] — Cox model stratified by IPSS-R score as per IRT

7. Secondary Outcome: Response Rate of Complete Remission (CR)/Marrow Complete Remission (mCR)/Partial Remission (PR)/Hematopoietic Improvement (HI))
Description: Percentage of complete remission (CR)/marrow Complete Remission (mCR)/partial remission (PR) & Hematological improvement (HI) as per investigator assessment according to IWG-MDS. CR: where the Bone marrow: ≤ 5% blasts with normal maturation of all cell lineages and Peripheral blood: where Hgb ≥ 10 g/dL AND Platelets ≥ 100*109/L AND Neutrophils ≥ 1.0*109/L AND Peripheral blasts 0%. mCR: where the Bone marrow ≤5% blasts and blast count decrease by ≥50% compared to baseline with or without improved blood counts or with or without transfusions. PR: All CR criteria except bone marrow: ≥50% decrease from baseline in blasts in bone marrow AND blast count in bone marrow >5%. HI: restoration or enhancement of the function of the body's blood cell-producing system that must last as least 8 weeks. HI definition is based on modified Hematological Improvement per IWG-MDS criteria in MDS & is the combination of Erythroid response (HI-E), Platelet response (HI-P) & Neutrophil response (HI-N).
Time Frame: approx. 32 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
Percentage of participants | 67.7 [54.9 to 78.8] | 61.3 [48.1 to 73.4]

8. Secondary Outcome: Duration of Complete Remission
Description: Duration of complete response is the time from the date of the first documented CR to the date of first documented relapse from CR or death due to any cause, whichever occurs first.
Time Frame: approx. 48 months
Population: Full Analysis Set (FAS): All randomized participants were included in the FAS (intent-to-treat population). Participant data in the FAS were analyzed according to the treatment and stratum they were assigned to when they were randomized. Analysis was done on participants who experienced a complete remission.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 15 | 13
Months | 17.97 [10.87 to 27.17] | 9.23 [5.09 to 17.97]
Statistical Analysis 1: Comparison: MBG453 + Hypomethylating Agents (HMA) vs Placebo + Hypomethylating Agents (HMA); Test type: Superiority; Hazard Ratio (HR) = 0.664, 95% CI 2-sided [0.240 to 1.838] — Cox model stratified by IPSS-R score as per IRT

9. Secondary Outcome: Time to Complete Remission
Description: Time from randomization to the first documented CR
Time Frame: Average of 7 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
Months | NA [NA to NA] — NA: Not estimable as there were insufficient number of participants with events. | NA [NA to NA] — NA: Not estimable as there were insufficient number of participants with events.
Statistical Analysis 1: Comparison: MBG453 + Hypomethylating Agents (HMA) vs Placebo + Hypomethylating Agents (HMA); Test type: Superiority; Hazard Ratio (HR) = 1.237, 95% CI 2-sided [0.588 to 2.601] — Cox model stratified by IPSS-R score as per IRT

10. Secondary Outcome: Percent of Participants Who Are Red Blood Cells (RBC)/Platelets Transfusion Independent After Randomization as Per IWG-MDS
Description: Improvement in RBC/platelets transfusion independence. RBC/platelets transfusion independence rate is defined as the percentage of participants having received no RBC/platelets transfusions during at least 8 consecutive weeks after randomization.
Time Frame: approx. 48 months
Population: Full Analysis Set (FAS): All randomized subjects were included in the FAS (intent-to-treat population). Participant data in the FAS were analyzed according to the treatment and stratum they were assigned to when they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
Percentage of participants
  Red blood cells (RBC) | 60.0 [47.1 to 72.0] | 64.5 [51.3 to 76.3]
  Platelets | 73.8 [61.5 to 84.0] | 74.2 [61.5 to 84.5]

11. Secondary Outcome: Red Blood Cells (RBC) Transfusion Independence Duration After Randomization
Description: The total duration of all transfusion independence periods is the sum of each period of the transfusion independence.
  RBC transfusions independence period is defined as the period for which participants having received no RBC transfusions during at least 8 consecutive weeks after randomization.
Time Frame: approx. 48 months
Population: Full Analysis Set (FAS): All randomized subjects were included in the FAS (intent-to-treat population). Participant data in the FAS were analyzed according to the treatment and stratum they were assigned to when they were randomized. Analysis done only on participants with at least one period of RBC transfusion independence post-baseline.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 39 | 40
Weeks | 46.29 [22.86 to 113.00] | 36.71 [20.29 to 65.36]

12. Secondary Outcome: Platelets Transfusion Independence Duration After Randomization
Description: The total duration of all transfusion independence periods is the sum of each period of the transfusion independence.
  Platelets transfusions independence period is defined as the period for which participants having received no platelets transfusions during at least 8 consecutive weeks after randomization.
Time Frame: approx. 48 months
Population: Full Analysis Set (FAS): All randomized participants were included in the FAS (intent-to-treat population). Participant data in the FAS were analyzed according to the treatment and stratum they were assigned to when they were randomized. Analysis done only on participants with at least one period of platelets transfusion independence post-baseline.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 48 | 46
Weeks | 44.36 [22.29 to 107.43] | 45.29 [25.14 to 80.00]

13. Secondary Outcome: Serum Concentrations for MBG453
Description: Pharmacokinetics (PK) of MBG453 when given in combination with hypomethylating agents (HMA)
Time Frame: 0hr pre-dose on Day 8 of each cycle until cycle 6 and on Day 8 of cycles 9, 12, 18 and 24, 2hr post-dose on Day 8 of C1 and C3, EOT (approx. 48 months) and up to 150 day of the safety follow up period; 1 cycle = 28 days
Population: Pharmacokinetic analysis set (PAS) included all participants in the Safety Set in the MBG453 arm only, who had at least one evaluable PK concentration.
Measure: Mean (Standard Deviation); unit: micro gram/mL
Arm/Group | MBG453 + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 49
micro gram/mL
  Cycle (C) 1 Day (D) 8 at 0 hour (hr) (pre-dose): number analyzed (Participants) | 47
  Cycle (C) 1 Day (D) 8 at 0 hour (hr) (pre-dose) | 0 (0)
  C1 D8 at 2 hr: number analyzed (Participants) | 37
  C1 D8 at 2 hr | 103 (72.4)
  C2 D8 at 0 hr (pre-dose): number analyzed (Participants) | 43
  C2 D8 at 0 hr (pre-dose) | 38.8 (20.5)
  C3 D8 at 0 hr (pre-dose) | 57.5 (32.1)
  C3 D8 at 2 hr: number analyzed (Participants) | 44
  C3 D8 at 2 hr | 149 (49.6)
  C4 D8 at 0 hr (pre-dose): number analyzed (Participants) | 42
  C4 D8 at 0 hr (pre-dose) | 70.7 (37.6)
  C5 D8 at 0 hr (pre-dose): number analyzed (Participants) | 42
  C5 D8 at 0 hr (pre-dose) | 76.7 (38.4)
  C6 D8 at 0 hr (pre-dose): number analyzed (Participants) | 39
  C6 D8 at 0 hr (pre-dose) | 85.0 (37.7)
  C9 D8 at 0 hr (pre-dose): number analyzed (Participants) | 30
  C9 D8 at 0 hr (pre-dose) | 97.3 (49.3)
  C12 D8 at 0 hr (pre-dose): number analyzed (Participants) | 22
  C12 D8 at 0 hr (pre-dose) | 103 (43.0)
  C18 D8 at 0 hr (pre-dose): number analyzed (Participants) | 11
  C18 D8 at 0 hr (pre-dose) | 97.7 (42.4)
  C24 D8 at 0 hr (pre-dose): number analyzed (Participants) | 4
  C24 D8 at 0 hr (pre-dose) | 134 (39.3)
  End of treatment (EOT): number analyzed (Participants) | 40
  End of treatment (EOT) | 50.0 (43.8)
  30 D Safety follow-up (f/u): number analyzed (Participants) | 11
  30 D Safety follow-up (f/u) | 44.4 (46.6)
  150 D Safety f/u: number analyzed (Participants) | 5
  150 D Safety f/u | 0 (0)

14. Secondary Outcome: Immunogenicity (IG) of MBG453 When Given in Combination of Hypomethylating Agents: ADA Prevalence
Description: Number of participants with at least one sample meeting the criteria at baseline. Anti-drug Antibody (ADA) prevalence equals ADA-positive at baseline.
Time Frame: at baseline
Population: The immunogenicity prevalence set included all participants in the full analysis set with a determinant baseline IG sample.
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 61
Participants | 11

15. Secondary Outcome: Immunogenicity of MBG453 When Given in Combination of Hypomethylating Agents: ADA-positive Participants
Description: Anti-drug Antibody (ADA) positive participants on-treatment was calculated as the number of participants with at least 1 on-treatment ADA-positive sample divided by the number of participants with a determinant baseline IG sample and at least one determinant post-baseline IG sample.
Time Frame: approx. 48 months
Population: Included all participants in the immunogenicity prevalence set with a determinant baseline IG sample and at least one determinant post-baseline IG sample.
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 60
Participants | 6

16. Post Hoc Outcome: All Collected Deaths
Description: Deaths were collected from randomization until end of trial, approx. 48 months.
Time Frame: from randomization until end of trial, approx. 48 months
Population: Clinical database population: All randomized participants: participants who died before treatment, during treatment and post-treatment.
Measure: Number; unit: Participants
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
Number analyzed (Participants) | 65 | 62
Participants
  Pre-treatment deaths | 0 | 1
  On-treatment deaths | 5 | 13
  Post-treatment deaths | 40 | 39
  Total deaths | 45 | 53

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the date of first administration of study treatment to 30 days after the date of the last administration of study treatment, up to maximum duration of 51.84 months (sabatolimab plus HMA) and 45.11 months (placebo + HMA). Deaths were collected from randomization until end of trial, approx. 48 months.
Description: Adverse Event: Any sign or symptom that occurs during the study treatment + 30 days post treatment.
Arm/Group | MBG453 + Hypomethylating Agents (HMA) | Placebo + Hypomethylating Agents (HMA)
All-Cause Mortality (participants affected / at risk) | 45/62 | 53/63
Serious Adverse Events (participants affected / at risk) | 38/62 | 43/63
Other Adverse Events (participants affected / at risk) | 61/62 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MBG453 + Hypomethylating Agents (HMA) (N=62) | Placebo + Hypomethylating Agents (HMA) (N=63)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 16 | 14
Hyperleukocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders and administration site conditions) | 1 | 0
Chills (General disorders and administration site conditions) | 0 | 1
Condition aggravated (General disorders and administration site conditions) | 0 | 1
Death (General disorders and administration site conditions) | 0 | 1
Disease progression (General disorders and administration site conditions) | 0 | 1
Fatigue (General disorders and administration site conditions) | 0 | 1
Gait disturbance (General disorders and administration site conditions) | 0 | 1
Pyrexia (General disorders and administration site conditions) | 1 | 9
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 3
Biliary sepsis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1
COVID-19 (Infections and infestations) | 2 | 2
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Dermo-hypodermitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2
Encephalitis (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 2
Gastrointestinal bacterial infection (Infections and infestations) | 1 | 0
Gingival abscess (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 9 | 11
Pneumonia fungal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 4 | 8
Septic shock (Infections and infestations) | 2 | 4
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MBG453 + Hypomethylating Agents (HMA) (N=62) | Placebo + Hypomethylating Agents (HMA) (N=63)
Anaemia (Blood and lymphatic system disorders) | 22 | 32
Febrile neutropenia (Blood and lymphatic system disorders) | 11 | 9
Neutropenia (Blood and lymphatic system disorders) | 25 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 13
Atrial fibrillation (Cardiac disorders) | 5 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 4
Conjunctival haemorrhage (Eye disorders) | 1 | 5
Abdominal distension (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 5
Constipation (Gastrointestinal disorders) | 29 | 26
Diarrhoea (Gastrointestinal disorders) | 27 | 15
Haemorrhoids (Gastrointestinal disorders) | 6 | 6
Nausea (Gastrointestinal disorders) | 15 | 19
Stomatitis (Gastrointestinal disorders) | 4 | 9
Toothache (Gastrointestinal disorders) | 4 | 2
Vomiting (Gastrointestinal disorders) | 7 | 6
Asthenia (General disorders and administration site conditions) | 11 | 7
Chest pain (General disorders and administration site conditions) | 2 | 4
Fatigue (General disorders and administration site conditions) | 14 | 8
Injection site erythema (General disorders and administration site conditions) | 2 | 4
Injection site reaction (General disorders and administration site conditions) | 4 | 10
Oedema (General disorders and administration site conditions) | 3 | 5
Oedema peripheral (General disorders and administration site conditions) | 8 | 7
Pain (General disorders and administration site conditions) | 3 | 4
Pyrexia (General disorders and administration site conditions) | 17 | 13
COVID-19 (Infections and infestations) | 9 | 4
Cellulitis (Infections and infestations) | 3 | 4
Nasopharyngitis (Infections and infestations) | 0 | 5
Oral herpes (Infections and infestations) | 3 | 6
Pneumonia (Infections and infestations) | 2 | 7
Respiratory tract infection (Infections and infestations) | 5 | 0
Urinary tract infection (Infections and infestations) | 9 | 3
Contusion (Injury, poisoning and procedural complications) | 6 | 0
Procedural pain (Injury, poisoning and procedural complications) | 4 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 5
Alanine aminotransferase increased (Investigations) | 4 | 12
Aspartate aminotransferase increased (Investigations) | 6 | 9
Blood alkaline phosphatase increased (Investigations) | 4 | 3
Blood bilirubin increased (Investigations) | 1 | 5
Blood creatinine increased (Investigations) | 2 | 5
Blood lactate dehydrogenase increased (Investigations) | 3 | 5
Gamma-glutamyltransferase increased (Investigations) | 2 | 7
Lymphocyte count decreased (Investigations) | 3 | 5
Neutrophil count decreased (Investigations) | 14 | 23
Platelet count decreased (Investigations) | 12 | 19
SARS-CoV-2 test negative (Investigations) | 5 | 7
Weight decreased (Investigations) | 10 | 8
White blood cell count decreased (Investigations) | 13 | 17
Decreased appetite (Metabolism and nutrition disorders) | 13 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 6
Dizziness (Nervous system disorders) | 8 | 5
Headache (Nervous system disorders) | 8 | 7
Paraesthesia (Nervous system disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 9 | 9
Acute kidney injury (Renal and urinary disorders) | 5 | 3
Dysuria (Renal and urinary disorders) | 4 | 3
Haematuria (Renal and urinary disorders) | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Erythema (Skin and subcutaneous tissue disorders) | 6 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 7
Purpura (Skin and subcutaneous tissue disorders) | 2 | 4
Rash (Skin and subcutaneous tissue disorders) | 12 | 8
Haematoma (Vascular disorders) | 4 | 3
Hypertension (Vascular disorders) | 7 | 7
Hypotension (Vascular disorders) | 3 | 6

LIMITATIONS AND CAVEATS:
A total of 127 subjects were randomized (65 to sabatolimab (S)+HMA arm, 62 to placebo (P)+HMA arm. However, only 125 subjects were treated (64 in S+HMA arm, 61 in P+HMA arm). Two subjects in S+HMA arm received only HMA, and, as a result, were reported in P+HMA arm in the safety dataset. Therefore, the safety dataset included a total of 62 subjects in the S+HMA arm & 63 subjects in the P+HMA arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e. data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03946670/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT03946670/SAP_001.pdf